CLINICAL TRIAL: NCT00115336
Title: Ketorolac Versus Ibuprofen for the Painful Crisis of Sickle Cell Disease - Southwestern Comprehensive Sickle Cell Center
Brief Title: Ketorolac Versus Ibuprofen to Treat Painful Episodes of Sickle Cell Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 191; U54HL070588 (NIH)
Record Dates: First submitted 2005-06-21; First posted 2005-06-22 (Estimated); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Hematologic Diseases; Anemia, Sickle Cell
Keywords: Blood Diseases; Sickle Cell Anemia
MeSH Terms: conditions — Hematologic Diseases; Anemia, Sickle Cell | interventions — Ketorolac Tromethamine; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1-Intravenous ketorolac and oral placebo (Active Comparator): Intravenous ketorolac and oral placebo
  Interventions: Drug: Intravenous Ketorolac
- 2-Intravenous placebo and oral ibuprofen (Active Comparator): Intravenous placebo and oral ibuprofen
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Intravenous Ketorolac — Intravenous ketorolac
  Other Names: Toradol
  Arms: 1-Intravenous ketorolac and oral placebo
Drug: Ibuprofen — Ibuprofen, taken orally
  Other Names: Motrin, Advil
  Arms: 2-Intravenous placebo and oral ibuprofen

SUMMARY:
The purpose of this study is to compare ketorolac, a potent, non-steroidal anti-inflammatory drug (NSAID), with ibuprofen, a commonly used NSAID, for the treatment of the painful crisis of sickle cell disease (SCD).

DETAILED DESCRIPTION:
BACKGROUND:

SCD is a common disorder among African Americans and other minority groups. It is characterized by chronic anemia and episodic vaso-occlusive crises. The most common of these crises is the painful crisis. Current treatment of the painful crisis includes rest, hydration, and analgesic medication. Morphine is the most commonly prescribed analgesic medication for moderate to severe painful episodes, but there are several side effects associated with its use, including somnolence, respiratory depression, constipation, dysphoria, and pruritus. Other analgesic medications, including NSAIDs, may improve pain control and decrease the need for morphine and other opioid drugs; however, more research is needed to confirm the benefits in individuals with SCD.

DESIGN NARRATIVE:

This study will enroll 120 children who will receive standard opioid and supportive therapy. In addition to this care, participants will be randomly assigned to receive one of the following: 1) intravenous ketorolac and oral placebo; or 2) intravenous placebo and oral ibuprofen. Outcome assessments will include the duration of hospitalization for opioid therapy; the degree of pain intensity and relief determined by validated pain scales; and the utilization of opioid medications during hospitalization. All participants will be monitored for potential adverse effects of the study medications by laboratory measurements and clinical assessments. Additionally, participants will self-report pain levels using the Oucher pain scale. Participants will be monitored for the development of adverse events, including gastrointestinal symptoms and deterioration of kidney function, as determined by daily kidney function tests including BUN, creatinine, and hematuria.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of any form of SCD, including sickle cell anemia, sickle-hemoglobin C disease, and sickle-ß˖ or ß°-thalassemia
* Currently experiencing an acute painful episode (vaso-occlusive crisis), defined as acute pain in the extremities, back, abdomen, or chest that has lasted at least 4 hours and is presumed to be due to SCD, with no other identified cause
* Onset of severe pain in its current location(s) must have occurred within 72 hours of study entry
* Intensity of pain must be great enough to necessitate hospitalization for opioid analgesia (e.g., failure of home and outpatient therapy)
* Ability to comprehend and use patient-controlled analgesia (PCA)
* Score of 6 or greater on the baseline pain scale

Exclusion Criteria:

* Temperature greater than or equal to 38.5ºC at the time of study entry or in the preceding 12 hours
* Has a new lobar pulmonary infiltrate or a diagnosis of acute chest syndrome (i.e., a new lobar pulmonary infiltrate and two or more of the following: temperature greater than 38ºC, tachypnea, dyspnea, intercostal or supraclavicular retractions, nasal flaring, chest wall pain, and an oxygen saturation of less than 90% in room air by pulse oximetry)
* Diagnosis of acute splenic or hepatic sequestration crisis (i.e., liver or spleen enlarged from steady-state size and Hgb level decreased 2 g/dL or more from steady-state value)
* Currently experiencing priapism
* Pain caused by suspected or confirmed hepatobiliary disease (e.g., cholecystitis or cholelithiasis)
* Chronic pain caused by suspected or confirmed aseptic or avascular necrosis of the femoral or humeral heads
* Chronic pain syndrome characterized by opioid tolerance and defined by hospitalization for at least 30 days for the management of pain in a 1 year period prior to study entry
* Current participation (last transfusion given within the 2 months prior to study entry) in a program of chronic transfusions for the management of SCD; the use of hydroxyurea alone is permitted
* Allergy or history of anaphylactoid reactions to aspirin or other NSAIDs
* Kidney dysfunction (i.e., serum creatinine concentration greater than 1.5 times the upper limit of normal for age)
* History of gastrointestinal bleeding or ulceration requiring medical therapy
* Concomitant bleeding disorder (e.g., von Willebrand disease, hemophilia, or a qualitative platelet defect)
* Any other medical condition that would make it unsafe to receive NSAIDs, as determined by the study physician
* PCA not preferred
* Use of ketorolac in the 30 days prior to study entry
* Use of scheduled (e.g., "around the clock") opioid analgesics in the 5 days before the onset of current acute painful crisis
* Pregnant

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2005-01; Primary Completion 2008-08 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles T. Quinn, MD, Study Chair — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Planned enrollment for the trial was 120 subjects. Accrual was extremely slow; only 10 participants were randomized before the trial was closed in 2008 due to lack of accrual. Less than 10% of planned enrollment was achieved.
Groups:
- IV Ketorolac / Oral Placebo: Intravenous ketorolac and oral placebo
- IV Placebo / Oral Ibuprofen: Intravenous placebo and oral ibuprofen
Period: Overall Study
Arm/Group | IV Ketorolac / Oral Placebo | IV Placebo / Oral Ibuprofen
Started | 6 | 4
Completed | 6 | 3
Not Completed | 0 | 1
Not completed — Hospital discharge before study drug | 0 | 1

BASELINE CHARACTERISTICS:
Population: One participant was randomized but was discharged (unexpectedly early) from the hospital before study drug was administered. Thus, no primary or secondary outcome data are available for this one participant.
Groups:
- IV Placebo / Oral Ibuprofen: Intravenous placebo abd oral ibuprofen
- Total: Total of all reporting groups
Arm/Group | IV Ketorolac / Oral Placebo | IV Placebo / Oral Ibuprofen | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 4 | 7
  Between 18 and 65 years | 3 | 0 | 3
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 15.4 [14.0 to 17.3] | 17.7 [15.6 to 18.2] | 16.7 [14.0 to 18.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Time to a 50% Reduction in Reported Pain Intensity
Description: The primary endpoint is the time to a 50% reduction in reported pain intensity. This endpoint is relative to the baseline pain intensity rating on the Oucher scale (minimum 0, maximum 10; higher scores indicate greater pain). The endpoint will be reached when the reported pain intensity is at least one-half of the baseline value on two consecutive measurements at least 4 hours apart. The time ascribed to the endpoint will be the time of the second of these two consecutive pain scales. Participants who do not have a 50% reduction in reported pain intensity, as defined above, before discharge from the hospital will be censored at the time of last rating on the Oucher pain scale before discharge from the hospital
Time Frame: Measured every 4 hours during hospitalization, over a mean hospitalization duration of 81.5 hours.
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | IV Ketorolac / Oral Placebo | IV Placebo / Oral Ibuprofen
Number analyzed (Participants) | 6 | 3
hours | 58.4 [29.3 to 87.4] | 68.0 [20.3 to 115.8]

2. Secondary Outcome: Duration of Hospitalization
Description: Time between admission to the hospital and discharge from the hospital
Time Frame: The duration of the entire hospitalization, over a mean hospitalization duration of 81.5 hours.
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | IV Ketorolac / Oral Placebo | IV Placebo / Oral Ibuprofen
Number analyzed (Participants) | 6 | 3
hours | 80.7 [19.3 to 142.1] | 83.0 [27.2 to 138.7]

3. Secondary Outcome: Total Parenteral Opioid Usage
Description: Sum of all parenteral opioids used during the study period in milligrams (mg) of morphine or morphine equivalents.
Time Frame: The duration of the entire hospitalization, over a mean hospitalization duration of 81.5 hours.
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: milligrams (mg) of morphine equivalents
Arm/Group | IV Ketorolac / Oral Placebo | IV Placebo / Oral Ibuprofen
Number analyzed (Participants) | 6 | 3
milligrams (mg) of morphine equivalents | 225.2 [17.0 to 433.3] | 264.6 [0 to 530.8]

4. Secondary Outcome: Occurrence of Azotemia
Description: Participants who had measured values of blood urea nitrogen (BUN), serum creatinine, or both that were above the upper limit of normal for age.
Time Frame: The duration of the entire hospitalization, over a mean hospitalization duration of 81.5 hours.
Population: Extremely slow accrual led to the trial closing in 2008. Because only 10% of planned enrollment was achieved, no analysis of the primary or secondary outcome data was performed because of lack of power and generalizability.
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ketorolac / Oral Placebo | IV Placebo / Oral Ibuprofen
Number analyzed (Participants) | 6 | 3
Participants | 0 | 0

5. Secondary Outcome: Fluid Retention
Description: Number of participants who had clinically overt fluid retention as determined by history, physical examination, vital signs, and weight (e.g., peripheral edema, increase in weight)
Time Frame: The entire study period (daily assessments during hospitalization [mean of 81.5 hours] and once at the 30-day follow-up visit, over a mean of 33.4 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Intravenous Ketorolac and Oral Placebo: Intravenous ketorolac and oral placebo
  Intravenous Ketorolac: Intravenous ketorolac
- Intravenous Placebo and Oral Ibuprofen: Intravenous placebo and oral ibuprofen
  Ibuprofen: Ibuprofen, taken orally
Arm/Group | Intravenous Ketorolac and Oral Placebo | Intravenous Placebo and Oral Ibuprofen
Number analyzed (Participants) | 6 | 3
Participants | 0 | 0

6. Secondary Outcome: Hematuria
Description: Number of participants who had microscopic hematuria as determined by urinalysis
Time Frame: The duration of the entire hospitalization, over a mean hospitalization duration of 81.5 hours.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ketorolac / Oral Placebo | IV Placebo / Oral Ibuprofen
Number analyzed (Participants) | 6 | 3
Participants | 4 | 1

7. Secondary Outcome: Dyspepsia
Description: Number of participants who reported discomfort in the stomach related to eating or drinking
Time Frame: as for outcome 5
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ketorolac / Oral Placebo | IV Placebo / Oral Ibuprofen
Number analyzed (Participants) | 6 | 3
Participants | 0 | 0

8. Secondary Outcome: Gastrointestinal Ulceration
Description: Number of participants who had gastrointestinal ulceration.
Time Frame: as for outcome 5
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ketorolac / Oral Placebo | IV Placebo / Oral Ibuprofen
Number analyzed (Participants) | 6 | 3
Participants | 0 | 0

9. Secondary Outcome: Bleeding
Description: Number of participants who had clinically overt bleeding from any site. This excludes microscopic hematuria only.
Time Frame: as for outcome 5
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ketorolac / Oral Placebo | IV Placebo / Oral Ibuprofen
Number analyzed (Participants) | 6 | 3
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Description: All adverse events were systematically assessed at all study visits according to the study protocol by trained study personnel. Adverse events were recorded for up to 30 days from discharge from the hospital.
Arm/Group | IV Ketorolac / Oral Placebo | IV Placebo / Oral Ibuprofen
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 6/6 | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Ketorolac / Oral Placebo (N=6) | IV Placebo / Oral Ibuprofen (N=4)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Fever (Immune system disorders) | 1 (1) | 1 (1)
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Extremely slow accrual led to the trial closing in 2008. Because less than 10% of planned enrollment was achieved, no statistical analysis of the primary or secondary outcome data was performed because of lack of power and generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No